CLINICAL TRIAL: NCT01812616
Title: A Two Part Study to Assess the Tolerability, Safety and Pharmacodynamics of Sativex in Combination With Dose-intense Temozolomide in Patients With Recurrent Glioblastoma
Brief Title: A Safety Study of Sativex Compared With Placebo (Both With Dose-intense Temozolomide) in Recurrent Glioblastoma Patients
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Jazz Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: GWCA1208 Part B
Record Dates: First submitted 2013-03-14; First posted 2013-03-18 (Estimated); Last update posted 2022-12-20 (Actual); Status verified 2022-12

CONDITIONS: Cancer
Keywords: Cancer; Safety
MeSH Terms: conditions — Neoplasms | interventions — nabiximols

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Sativex and Dose-Intense Temozolomide (Experimental): Patients will received Sativex and Dose-Intense Temozolomide in a double-blind manner
  Interventions: Drug: Sativex
- Placebo and Dose-Intense Temozolomide (Placebo Comparator): Patients will received placebo and Dose-Intense Temozolomide and in double-blind manner
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Sativex — Administered orally as a spray to the cheek according to a standard dose titration regimen, until patients reach a maximum tolerated dose (maximum 12 sprays per day). Each spray delivers 100 μl (Δ9tetrahydrocannabinol (THC), 27 mg/ml: Cannabidiol (CBD), 25 mg/ml).
  Other Names: THC/CBD spray; Nabiximols; GW-1000-02
  Arms: Sativex and Dose-Intense Temozolomide
Drug: Placebo — Administered orally as a spray to the cheek according to a standard dose titration regimen, until patients reach a maximum tolerated dose (maximum 12 sprays per day). Each spray delivers 100 μl ethanol:propylene glycol (50:50) excipients, with peppermint oil (0.05%) flavouring and Food, Drugs & Cosmetics (FD&C)certified color additives; FD&C Yellow No.5 (E102 tartrazine) (0.0260%), FD&C Yellow No.6 (E110 sunset yellow) (0.0038%), FD&C Red No. 40 (E129 Allura red AC) (0.00330%) and FD&C Blue No.1 (E133 Brilliant blue FCF) (0.00058%).
  Other Names: Placebo comparator
  Arms: Placebo and Dose-Intense Temozolomide

SUMMARY:
An open-label phase to assess the frequency and severity of adverse events in recurrent glioblastoma patients receiving Sativex in combination with dose-intense Temozolomide (Part A). A randomisation phase to assess the safety of Sativex compared with placebo (Part B). Part B will be reported here.

DETAILED DESCRIPTION:
Patients will receive Sativex and dose-intense Temozolomide in an open-label phase. The incidence of adverse events will be monitored (Part A). An investigator led Safety Review Team will assess the safety profile of the open-label patients and decide whether the study can progress to the randomisation phase (Part B). Patients who enrol in the randomisation phase patients will receive either Sativex or placebo. The safety of Sativex compared to placebo will be assessed by pharmacokinetic analysis of Temozolomide and its metabolites, clinical laboratory tests, adverse events and vital signs.

ELIGIBILITY:
Inclusion Criteria:

* Patient is willing and able to give informed consent for participation in the study.
* Patient is aged 18 years or above.
* Histopathologically confirmed diagnosis of grade four Glioblastoma Multiforme as per World Health Organisation classification.
* Evidence of patients first tumour progression (as determined by Revised Assessment in Neuro-Oncology) following radiation and first line chemotherapy with Temozolomide.
* If taking steroids, then the dose must be stable or decreasing.
* Karnofsky performance scale of 60% or greater.
* Patient is able (in the investigators opinion) and willing to comply with all study requirements.
* Patient is willing for his or her name to be notified to the responsible authorities for participation in this study, as applicable in individual countries.
* Patient is willing to allow his or her primary care practitioner and consultant, if appropriate, to be notified of participation in the study.

Exclusion Criteria:

* Patients with Glioblastoma Multiforme secondary to low-grade glioma or anaplastic glioma (anaplastic astrocytoma or anaplastic oligodendroglioma).
* Patients currently receiving treatment for recurrent Glioblastoma Multiforme.
* Less than a four week interval since prior chemotherapy.
* Less than a 12 week interval since prior radiotherapy unless there is either: a) histopathology confirmation of recurrent tumour, or b) new enhancement on Magnetic Resonance Imaging outside of the radiotherapy treatment field.
* Presence of extra-cranial metastatic disease.
* Any surgery, including intracranial biopsy (not including minor diagnostic procedures such as lymph node biopsy) within two weeks of baseline disease assessments; or not fully recovered from any side effects of previous procedures.
* Any history of a different malignancy unless the patient has remained disease-free for at least three years and are at low risk for recurrence of that malignancy (cervical cancer in situ, and basal cell or squamous cell carcinoma of the skin are exempt from this criterion if treatment has occurred).
* Have previously received first line chemotherapy other than Temozolomide.
* Presents with Leptomeningeal dissemination.
* Have previously received stereotactic radiotherapy, convection enhanced delivery or brachytherapy (as gliosis/scarring from these modalities may limit delivery).
* The patient is currently using or has used cannabis or cannabinoid based medications within 30 days of study entry and is unwilling to abstain for the duration of the study.
* Any known or suspected history of a substance abuse/dependence disorder, current heavy alcohol consumption (>60g of pure alcohol per day for men, >40 g of pure alcohol per day for women), current use of an illicit drug or current non prescribed use of any prescription drug.
* Any history or immediate family history of schizophrenia, other psychotic illness, severe personality disorder or other significant psychiatric disorder other than depression associated with their underlying condition.
* Has experienced myocardial infarction or clinically significant dysfunction within the last 12 months or has a cardiac disorder that, in the opinion of the investigator would put the patient at risk of clinically significant arrhythmia or myocardial infarction.
* Has grade 3 or above toxicity by Common Terminology Criteria for Adverse Events criteria.
* Female patients of child bearing potential and male patients whose partner is of child bearing potential, unless willing to ensure that they or their partner use effective contraception, for example, oral contraception, double barrier, intra-uterine device, during the study and for three months thereafter (however a male condom should not be used in conjunction with a female condom).
* Female patients who are pregnant, lactating or planning pregnancy during the course of the study and for three months thereafter.
* Patient who have received an Investigational Medicinal Product within the four weeks prior to the screening visit.
* Any other significant disease or disorder which, in the opinion of the investigator, may either put the patient at risk because of participation in the study, or may influence the result of the study, or the patient's ability to participate in the study.
* Travel outside the country of residence planned during the study.
* Patients previously enrolled into this study and received either Investigational Medicinal Product or Dose-Intense Temozolomide.
* Any known or suspected hypersensitivity to cannabinoids or any of the excipients of the Investigational Medicinal Product.
* Any known allergy to or other intolerability to Temozolomide.
* Following a physical examination, the patient has any abnormalities that, in the opinion of the investigator would prevent the patient from safe participation in the study.
* Unwilling to abstain from donation of blood during the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 21 (Actual)
Dates: Start 2014-09; Primary Completion 2016-06 (Actual); Study Completion 2016-06 (Actual)

PRIMARY OUTCOMES:
Incidence of Adverse Events as a Measure of Patient Safety. | Study Day 1 - Day 358
  Adverse events will be coded according to the current medical dictionary for regular activities graded using the Common Terminology Criteria for Adverse Events criteria. The number of patients who experienced an adverse event whilst on treatment will be presented.

SECONDARY OUTCOMES:
The number of patients with Progression Free Survival at six months (PFS6) | Study Day 1 - Day 190
  PFS6 will be assessment at Visit 11 (Day 190). Progression of disease will be determined from Response Assessment in Neuro-Oncology tumour assessment (based on Magnetic Resonance Imaging scans). The number of patients with PFS6 will be presented for the individual treatment groups.
Overall Survival | Study Day 1 - Day 358
  Overall survival will be assessed at the end of the treatment visit (Day 358 or at early termination). The number of surviving patients in each group from the randomisation phase (Part B) will be presented.

CONTACTS AND LOCATIONS:
Locations (11):
- Germany (4):
  - Klinik für Onkologie, Hämatologie und Stammzelltransplantation, Universitätsklinikum Aachen RWTH, Aachen
  - Neurologie des Klinikums Altenburger Land, Altenburg
  - Zentrum für Neuroonkologie der Universität Duesseldorf, Düsseldorf
  - Strahlenklinik der Universität Erlangen, Erlangen
- United Kingdom (7):
  - The Clatterbridge Cancer Centre NHS Foundation Trust, Bebington, Wirral
  - St James's Institute of Oncology, St James's University Hospital, Leeds, Yorkshire
  - Bristol Haematology & Oncology Centre, Bristol
  - Queen's Centre for Haematology & Oncology, Castle Hill Hospital, Cottingham
  - West of Scotland Beatson Cancer Centre, Glasgow
  - Guy's & St Thomas' NHS Foundation Trust, of St Thomas' Hospital, London
  - The Christie NHS Foundation Trust, Manchester

REFERENCES:
- [Derived] Twelves C, Sabel M, Checketts D, Miller S, Tayo B, Jove M, Brazil L, Short SC; GWCA1208 study group. A phase 1b randomised, placebo-controlled trial of nabiximols cannabinoid oromucosal spray with temozolomide in patients with recurrent glioblastoma. Br J Cancer. 2021 Apr;124(8):1379-1387. doi: 10.1038/s41416-021-01259-3. Epub 2021 Feb 24. PMID 33623076